CLINICAL TRIAL: NCT01617070
Title: Pilot Study to Evaluate Melatonin Secretion as a Marker of Decreased Serotonin in Individuals With PKU: Evaluation of the CNS Effects of Tetrahydrobiopterin
Brief Title: Effects of Kuvan on Melatonin Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Shoji Yano, M.D., Ph.D, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USC Kuvan Melatonin
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Phenylketonuria (PKU)
Keywords: Tetrahydrobiopterin; Kuvan; Phenylketonuria (PKU); Large Neutral Amino Acids; Serotonin; Dopamine; Melatonin
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LNAA, washout, Kuvan, and LNAA+Kuvan (Experimental): One group of 12 subjects, each under 4 conditions (each phase is 4 weeks)
  Interventions: Drug: Kuvan; Dietary Supplement: Large Neutral Amino Acid Therapy

INTERVENTIONS:
Drug: Kuvan — Dosed at 20 mg/kg; PO; Phase 3, Phase 4
  Other Names: Tetrahydrobiopterin
Dietary Supplement: Large Neutral Amino Acid Therapy — Dosed by weight: weight x .5 = total tablets per day; PO; Phase 1, Phase 4; taken with food
  Other Names: LNAA

SUMMARY:
This study examines the effect of tetrahydrobiopterin (Kuvan) and Large Neutral Amino Acid (LNAA) therapy on melatonin and dopamine levels in individuals with Phenylketonuria (PKU). The investigators hypothesize that Kuvan therapy will improve melatonin secretion and urine dopamine levels to some extent. However significantly greater responses in melatonin and dopamine secretions may be observed with combined treatment with Kuvan and supplementation of LNAA.

DETAILED DESCRIPTION:
Background: Phenylketonuria (PKU) is a genetic condition due to missing one of the key enzymes of phenylalanine (Phe) degradation. The missing enzyme is phenylalanine hydroxylase (PAH). Because of the deficiency of the enzyme, plasma Phe is highly elevated compared with other plasma amino acids. This abnormal ratio i.e., Phe vs. each of the other large neutral amino acids (LNAA) which are transported into the brain as precursors of neurotransmitters through the common transporter LAT1, is likely to contribute to neurotransmitter deficiencies in individuals with PKU. Patients who do not restrict Phe intake develop mental retardation and neuropsychological disorders. Treatment of PKU has been historically limited to restriction of Phe intake, meaning protein restriction.

The FDA recently approved a new medication, Kuvan, a synthetic form of tetrahydrobiopterin (BH4) manufactured by BioMarin Pharmaceutical Inc., for patients with PKU. Kuvan is a cofactor for PAH, tyrosine hydroxylase, and tryptophan hydroxylase. Patients with PKU typically undergo a month-long trial of Kuvan to determine if they are responders to the drug, meaning blood phenylalanine drops by more than 30 percent. Those who are not responders do not usually continue Kuvan, however our recent study (HS 08-00147) showed that classical PKU patients who are not Kuvan responders demonstrated improvement in their maladaptive behaviors, suggesting some effects of Kuvan in the CNS system without reducing blood phenylalanine concentrations (Moseley et al, manuscript under preparation). Seven subjects who did not respond to Kuvan with lower blood Phe levels had significant increases in blood tyrosine after 6 months (p=0.015), along with improvement in the Vineland Internalizing and Overall Maladaptive Behavior Indexes at 12 months (p=0.032 and 0.049, respectively). Kaufman reported that Kuvan at dose of 20 mg/kg/day increased CSF BH4 levels (1). Based on these observations, it is likely that Kuvan has some effects on neurotransmitter metabolism.

Supplementation of large neutral amino acids (LNAA) as a medical food has been used in Europe for the past 25 years and it is believed to be effective in treating patients with PKU. In the article by Shindeler et al. (2), 16 individuals (7 males and 9 females; age 11y to 45 y) participated in the study which consisted 4 weeks wash-out and 4 two-weeks stages (on phenylalanine restricted diet and with/without LNAA, and on no phenylalanine restricted diet and with/without LNAA). No specific adverse effects are reported in the article. Large neutral amino acid therapy for the treatment of PKU has been done in the past (3). LNAA is used primarily for adolescents and adults who cannot adhere to the standard phe-restricted diet. LNAA treatment has been approved for PKU patients just like other special formulas. Our previous studies have demonstrated deficiency of serotonin in the brain, as evidenced by low nocturnal melatonin secretion and reduced urine dopamine compared to controls, and that supplementation with LNAA improves, but does not normalize these markers.

Rationale: Patients with PKU are thought to be deficient in tyrosine and tryptophan in the brain tissue level because of the abnormal phe/tyrosine and phe/tryptophan ratios. Previous studies showed low serotonin levels in cerebrospinal fluid in PKU individuals and some improvement was observed after tryptophan supplementation (4). Our prior study suggested deficiency of tryptophan in the brain tissue was demonstrated by low nocturnal melatonin secretion and 6-sulfatoxymelatonin, which is a stable metabolite of melatonin (5). LNAA supplementation resulted in some improvement in melatonin secretion, however, melatonin secretion in patients with PKU on LNAA was still significantly lower than the control group. Supplementation of Kuvan may activate the brain tyrosine and tryptophan hydroxylases (6), resulting in improvement of nocturnal melatonin secretion and urine melatonin and dopamine concentrations. By supplementing LNAA increased amount of neurotransmitter precursor amino acids will be transported into the brain and activated brain tyrosine and tryptophan hydroxylases by Kuvan will act on these precursors to produce neurotransmitters, i.e., serotonin and dopamine. These synergistic effects may increase melatonin and dopamine levels to closer to the control levels.

Aims of the Study: To show scientific evidence of improvement in metabolism of neurotransmitters including serotonin and dopamine in patients with PKU treated with LNAA only, Kuvan only, and Kuvan and LNAA.

Objectives: This investigator initiated study has three objectives: (1) To evaluate if tetrahydrobiopterin (Kuvan) supplementation has beneficial effects on melatonin secretion and urine dopamine levels in individuals with PKU when they are and are not treated with large neutral amino acids; (2) To demonstrate synergistic effects of LNAA supplementation and Kuvan therapy in improvement of neurotransmitter metabolism in individuals with PKU; and (3) To gather pilot information necessary to design a larger, multicenter trial of these interventions, should results of these pilot studies indicate further study is warranted.

Study Methodology: This study will be conducted in adult patients with PKU in four 4-week phases: phase I (large neutral amino acid/LNAA), phase II (Washout), phase III (Kuvan only) and phase IV (Kuvan and LNAA). Kuvan supplementation will be adjusted to provide 20 mg/kg/day. LNAA therapy is adjusted to the manufacturer's instruction (total tablets of LNAA is 1/2 X BW kg). On the last day of each phase, subjects will stay approximately 14 to 18 hours overnight at the CTU at USC University Hospital. Blood specimens will be collected every 2 hours from 7:00 pm to 7:00 am. First void urine will be collected on the day of discharge (patients will be asked to void urine at 11:00 pm and the first void urine will be collected).

Blood will be collected in a red top tube (5 ml) through an IV line which is saline locked during the study period. Avoid hemolysis by collecting blood through an IV line into a reasonably large peripheral vein. Blood will be left to clot for 45 minutes at room temperature (18-28 C) and protected from light (a dim flash light or a yellow light < 100 lux). Serum will be collected and stored at - 20 C until they are subjected to analysis for plasma melatonin and plasma amino acids. Urine 20 ml first void sample will be collected into two plain tubes (10 ml per each tube) and stored in a deep freezer (-20 C) until subjected to be analyzed for dopamine and 6-sulfatoxymelatonin.

This is an open-labeled study. During all four 4-week phases, subjects will remain on their protein-restricted diet. LNAA tablets are not considered a medicine, but are under the category of medical foods; examples include low protein foods. LNAA tablets will be provided by the LNAA manufacture (Applied Nutrition). Kuvan will be taken per orally with breakfast and LNAA tablets will be taken with meals three times per day.

ELIGIBILITY:
Inclusion Criteria:

* Adult English-speaking patients who have confirmed PKU, and have tolerated Kuvan therapy at 20 mg/kg/day in the past, and are currently on the LNAA supplements will be considered as candidates for the study.
* Subjects must be able to stop LNAA therapy for 4 weeks.
* This will be determined by the subjects themselves, based on their past personal experiences.

Exclusion Criteria:

* Individuals who have never taken Kuvan, who have never been on LNAA therapy, who are under the age of 18, or who do not speak English will be excluded.
* Subjects who cannot stop LNAA therapy for 4 weeks will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Yano, M.D., Ph.D., Principal Investigator — USC Keck School of Medicine, Dept. of Pediatrics, Genetics Division
Locations (1):
- Keck School of Medicine, Clinical Trials Unit at Keck Medical Center of USC, Los Angeles, California, United States

REFERENCES:
- [Background] Kaufman S, Kapatos G, McInnes RR, Schulman JD, Rizzo WB. Use of tetrahydropterins in the treatment of hyperphenylalaninemia due to defective synthesis of tetrahydrobiopterin: evidence that peripherally administered tetrahydropterins enter the brain. Pediatrics. 1982 Sep;70(3):376-80. PMID 7110811
- [Background] Schindeler S, Ghosh-Jerath S, Thompson S, Rocca A, Joy P, Kemp A, Rae C, Green K, Wilcken B, Christodoulou J. The effects of large neutral amino acid supplements in PKU: an MRS and neuropsychological study. Mol Genet Metab. 2007 May;91(1):48-54. doi: 10.1016/j.ymgme.2007.02.002. Epub 2007 Mar 23. PMID 17368065
- [Background] Lou H. Large doses of tryptophan and tyrosine as potential therapeutic alternative to dietary phenylalanine restriction in phenylketonuria. Lancet. 1985 Jul 20;2(8447):150-1. doi: 10.1016/s0140-6736(85)90250-8. No abstract available. PMID 2862338
- [Background] Nielsen JB, Lou H, Güttler F. Effects of diet discontinuation and dietary tryptophan supplementation on neurotransmitter metabolism in phenylketonuria. Brain Dysfunction 1:51-56. 1988.
- [Background] Zimmermann RC, McDougle CJ, Schumacher M, Olcese J, Heninger GR, Price LH. Urinary 6-hydroxymelatonin sulfate as a measure of melatonin secretion during acute tryptophan depletion. Psychoneuroendocrinology. 1993;18(8):567-78. doi: 10.1016/0306-4530(93)90034-i. PMID 8127947
- [Background] Katz I, Lloyd T, Kaufman S. Studies on phenylalanine and tyrosine hydroxylation by rat brain tyrosine hydroxylase. Biochim Biophys Acta. 1976 Oct 11;445(3):567-78. doi: 10.1016/0005-2744(76)90111-x. PMID 9989
- [Result] Yano S, Moseley K, Fu X, Azen C. Evaluation of Tetrahydrobiopterin Therapy with Large Neutral Amino Acid Supplementation in Phenylketonuria: Effects on Potential Peripheral Biomarkers, Melatonin and Dopamine, for Brain Monoamine Neurotransmitters. PLoS One. 2016 Aug 11;11(8):e0160892. doi: 10.1371/journal.pone.0160892. eCollection 2016. PMID 27513937

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: LNAA, washout, Kuvan, and LNAA+Kuvan
  One group of 10 subjects, each under 4 conditions (each phase is 4 weeks)
  Kuvan: Dosed at 20 mg/kg; PO; Phase 3, Phase 4
  Large Neutral Amino Acid Therapy: Dosed by weight: weight x .5 = total tablets per day; PO; Phase 1, Phase 4; taken with food
Period: LNAA (4 Weeks)
Arm/Group | All Study Participants
Started | 10
Completed | 10
Not Completed | 0
Period: Washout (4 Weeks)
Arm/Group | All Study Participants
Started | 10
Completed | 10
Not Completed | 0
Period: BH4 Therapy (4 Weeks)
Arm/Group | All Study Participants
Started | 10
Completed | 10
Not Completed | 0
Period: BH4 and LNAA (4 Weeks)
Arm/Group | All Study Participants
Started | 10
Completed | 9
Not Completed | 1
Not completed — started medication interfere with study | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Serum Melatonin at the End of 4 Weeks
Description: Evaluated for each subject under 4 conditions (washout, LNAA only, Kuvan only and LNAA+Kuvan)
Time Frame: measured every 4 weeks up to 16 weeks
Population: Participates who completed all phases were measured.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- LNAA: LNAA
  Large Neutral Amino Acid Therapy: Dosed by weight: weight x .5 = total tablets per day; PO; Phase 1, Phase 4; taken with food
- Washout: no Kuvan or LNAA or any medical food products. Limited protein intake diet.
- BH4 (Kuvan): Kuvan (BH4): Dosed at 20 mg/kg; PO; Phase 3, Phase 4
- BH4 and LNAA: Kuvan: Dosed at 20 mg/kg; PO; Phase 3, Phase 4
  Large Neutral Amino Acid Therapy: Dosed by weight: weight x .5 = total tablets per day; PO; Phase 1, Phase 4; taken with food
Arm/Group | LNAA | Washout | BH4 (Kuvan) | BH4 and LNAA
Number analyzed (Participants) | 9 | 9 | 9 | 9
pg/ml | 266.9 (165.7) | 205.7 (133.1) | 220.4 (138.5) | 301.2 (179.4)

2. Primary Outcome: Urine 6-sulfatoxymelatonin at the End of 4 Weeks
Description: Evaluated for each subject under 4 conditions (washout, LNAA only, Kuvan only and LNAA+Kuvan)
Time Frame: measured every 4 weeks up to 16 weeks
Population: Participates who completed all phases were measured.
Measure: Mean (Standard Deviation); unit: ng/mg Creatinine
Arm/Group | LNAA | Washout | BH4 (Kuvan) | BH4 and LNAA
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng/mg Creatinine | 14.5 (9.0) | 8.2 (4.8) | 8.6 (5.7) | 13.2 (9.3)

3. Primary Outcome: Urine Dopamine at the End of 4 Weeks
Description: Evaluated for each subject under 4 conditions (washout, LNAA only, Kuvan only and LNAA+Kuvan)
Time Frame: measured every 4 weeks up to 16 weeks
Population: Participates who completed all phases were measured.
Measure: Mean (Standard Deviation); unit: ug/gCreatinine
Arm/Group | LNAA | Washout | BH4 (Kuvan) | BH4 and LNAA
Number analyzed (Participants) | 9 | 9 | 9 | 9
ug/gCreatinine | 63.7 (26.7) | 42.6 (19.3) | 46.0 (16.8) | 67.6 (28.4)

ADVERSE EVENTS:
Arm/Group | LNAA | Washout | BH4 (Kuvan) | BH4 and LNAA
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes